CLINICAL TRIAL: NCT01381211
Title: Transarterial RAdioembolization Versus ChemoEmbolization for the Treatment of HCC: A Multicenter Randomized Controlled Trial (TRACE Trial)
Brief Title: Transarterial RAdioembolization Versus ChemoEmbolization for the Treatment of Hepatocellular Carcinoma (HCC)
Acronym: TRACE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: based on interim analysis results
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/050
Record Dates: First submitted 2011-06-14; First posted 2011-06-27 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Intermediate stage hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yttrium-90 radioembolization (90Y-RE) (Active Comparator)
  Interventions: Drug: 90Y-RE
- Transarterial chemoembolization with drug eluting beads (Active Comparator): Transarterial chemoembolization is performed with drug eluting beads, polyvinyl alcohol-based microspheres (DC Beads, Biocompatibles) loaded with the chemotherapeutic agent doxorubicin.
  Interventions: Drug: TACE-DEB

INTERVENTIONS:
Drug: TACE-DEB — Transcatheter arterial chemoembolization (TACE) is performed with drug eluting beads (DEB), polyvinyl alcohol-based microspheres loaded with the chemotherapeutic agent doxorubicin.
  Arms: Transarterial chemoembolization with drug eluting beads
Drug: 90Y-RE — Glass Yttrium-90 microspheres (TheraSphere®; MDS Nordion Inc.) will be used
  Arms: Yttrium-90 radioembolization (90Y-RE)

SUMMARY:
Hepatocellular carcinoma (HCC) is a primary malignant tumor of the liver that accounts for an important health problem worldwide. In only 10% - 15% of all patients with HCC, tumors are considered resectable at presentation. In contrast to metastatic liver disease, there is no role for systemic chemotherapy in the treatment of HCC. Today only evidence is available for Sorafenib, a tyrosine kinase inhibiting agent. The arsenal of non-surgical therapies can roughly be divided into local ablative, transarterial and systemic therapies. In well selected patients, local ablative therapy can offer favorable long term results.

For patients with disease confined to the liver, but locally more advanced, transarterial treatment modalities are proposed. These therapies exploit the dual blood supply to the liver. HCC derives its blood supply almost entirely from the hepatic artery, while liver parenchyma derives > 75% of its blood supply from the portal vein. Antitumoral agents, such as cytotoxic drugs or radionuclides, can be delivered in close proximity of the tumor.

Examples of transarterial therapies are: transarterial chemoembolization (TACE), bland transarterial embolization (TAE), transarterial chemoembolization with drug eluting beads (TACE-DEB) and transarterial radioembolization with Iodine-131 or Yttrium-90.

TACE is currently the gold standard for treatment of patients with intermediate stage HCC, with a reported median survival of around 17 months. A novel development in the TACE treatment for HCC is the drug-eluting bead (DEB). Recently performed small clinical trials reported the efficacy of DEBs in the treatment of intermediate stage HCC, which is substantially higher compared to conventional TACE.

Yttrium-90 radioembolization (90Y-RE) is a relatively recently developed technique which implements transarterial administration of minimally embolic microspheres loaded with Yttrium-90, a β-emitting isotope, delivering selective internal radiation to the tumor.

In this study the investigators want to prospectively compare TACE-DEB and 90Y-RE, two novel treatments that both have theoretical and/or proven advantages compared to the use of conventional TACE, in patients with intermediate stage HCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* The diagnosis HCC is confirmed by typical appearance on imaging or cytohistological evaluation (liver biopsy).
* Accurate staging:

MRI of the liver CT-scan of the abdomen and thorax bone scintigraphy, only in case of clinical symptoms suggestive of skeletal metastases.

Exclusion Criteria:

* Hypersensitivity to doxorubicin
* Pregnancy or breastfeeding
* Age under 18 years
* Child-Pugh score >B7
* ECOG performance status (PST) > 1
* Bilirubin > 2.6 mg/dl
* AST/ALT >5x upper limit of normal (ULN)
* >50% of liver involvement
* Main portal vein (right, left or common trunk) thrombosis
* Extra-hepatic disease
* Previous treatment of study target lesions
* 99mTc-labelled macroaggregated albumin (99mTc-MAA) scintigraphy shows lack of MAA uptake in tumor (photopenic lesion)
* Activity > 610 MBq and activity reduction would imply a liver target dose > 80 Gy
* patients who are declared incompetent or suffering from physic disorders that make a comprehensive judgement impossible, such as psychosis.
* Unmanageable intolerance for contrast medium
* Life expectancy < 3 months or otherwise impossible follow-up
* Inadequate bone marrow, liver and/or renal function
* other contraindications to hepatic embolization procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Time to Progression (TTP). | Patients will be followed over a 2 years period.
  Tumor progression is defined according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST) response evaluation criteria. The mRECIST evaluation criteria define progressive disease by the implication of target lesions response, non-target lesions response and the occurrence of new lesions.

SECONDARY OUTCOMES:
Time to Local Progression (TLP). | Since start of treatment untill local tumor progression with a maximum of 2 years follow up.
  In both study arms, treatment is done selectively for the lesions within the perfusion area (may be lobar, segmental or subsegmental), as visualized with Cone-Beam CT prior to intervention.
Survival of patients dedicated to either treatment arm. | Patients are followed for up to 2 years.
  Survival of patients is followed.
Quality of life EQ5D | Before treatment and after treatment on a 3 monthly interval during 2 years.
  Quality of life as measured with The Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) scale, The Short Form (36) Health Survey, EuroQol Group 5-Dimension Self-Report Questionnaire score (EQ5D) and European Organization for Research and Treatment of Cancer Quality of Life (EORTC-QLQ30).
Tumor response to therapy according to mRECIST criteria | Before treatment and after treatment on a 3 monthly interval during 2 years.
  European Association for the Study of the Liver (EASL) response will be obtained based on the following: complete response, partial response, stable disease.
Treatment-related costs. | After follow up of 2 year.
  Treatment-related costs, in terms of cost of therapy and number of hospitalization days, in these patients.
Toxicities and adverse events (recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 3.0) | 6 months following last treatment
  The number of patients with AEs, SAEs and SUSARs and the total number of AEs, SAEs and SUSARs in both treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Defreyne, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Dhondt E, Lambert B, Hermie L, Huyck L, Vanlangenhove P, Geerts A, Verhelst X, Aerts M, Vanlander A, Berrevoet F, Troisi RI, Van Vlierberghe H, Defreyne L. 90Y Radioembolization versus Drug-eluting Bead Chemoembolization for Unresectable Hepatocellular Carcinoma: Results from the TRACE Phase II Randomized Controlled Trial. Radiology. 2022 Jun;303(3):699-710. doi: 10.1148/radiol.211806. Epub 2022 Mar 8. PMID 35258371
- [Derived] Seinstra BA, Defreyne L, Lambert B, Lam MG, Verkooijen HM, van Erpecum KJ, van Hoek B, van Erkel AR, Coenraad MJ, Al Younis I, van Vlierberghe H, van den Bosch MA. Transarterial radioembolization versus chemoembolization for the treatment of hepatocellular carcinoma (TRACE): study protocol for a randomized controlled trial. Trials. 2012 Aug 23;13:144. doi: 10.1186/1745-6215-13-144. PMID 22913492